CLINICAL TRIAL: NCT06068361
Title: Diagnostic Evaluation of Dementia with Lewy Bodies Using a Multimodal Approach: EEG, Cognitive, Biological and MRI Biomarkers
Brief Title: Diagnostic Evaluation of Dementia with Lewy Bodies Using a Multimodal Approach
Acronym: EEG-EDELY
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association des Aidants et Malades à Corps de Lewy (A2MCL) (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP231168; 2023-A00961-44 (Other: ID RCB number)
Record Dates: First submitted 2023-09-29; First posted 2023-10-05 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Lewy Bodies Disease; Alzheimer Disease; Cognitive Impairment
Keywords: EEG; MRI; Plasma biomarkers
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- DLB patients: Dementia with Lewy bodies according to the revised criteria of Mc Keith 2017
  Interventions: Diagnostic Test: EEG
- AD patients: Alzheimer's disease according to McKhann et al., 2011 criteria including CSF biomarkers (an abnormal level of beta-amyloid 1-42 protein [Ab42] or a pathological Ab42/Ab40 ratio and an abnormal level of phosphorylated tau [p-tau])
  Interventions: Diagnostic Test: EEG
- Control: Subjective cognitive complaint, with a normal brain MRI and neurological examination, without any elements in favor of a neurodegenerative disease
  Interventions: Diagnostic Test: EEG

INTERVENTIONS:
Diagnostic Test: EEG — 32-electrode EEG (resting state, passive auditory and active visual task) + simultaneous recording with a 4 dry electrode EEG cap

SUMMARY:
Dementia with Lewy body disease (DLB) is the second leading cause of degenerative cognitive disorder after Alzheimer's disease (AD). Its variable clinical expression makes diagnosis difficult. To date, there is no validated DLB diagnostic biomarker, despite several biomarkers in development (EEG, MRI, biology).

Studies have shown that an improvement in diagnostic performance could be obtained by combining different modalities biomarkers using machine learning.

The aim of this research is to identify the best combination of multimodal biomarkers for the diagnosis of DLB (EEG, MRI, biology, cognitive scores), using a machine learning approach applied to a clinical cohort.

DETAILED DESCRIPTION:
Study population: Observational prospective cohort study including over 24 months at the GHU AP-HP. Nord Lariboisière, Cognitive Neurology Center : 50 probable DLB patients, 50 AD patients, and 30 control subjects with subjective cognitive impairment but without any element in favor of neurodegenerative disorders. Total clinical dataset n= 130.

Act :

* 32-electrode EEG (resting state, passive auditory and active visual task).
* 4 dry electrode EEG cap simultaneously with the 32-electrode EEG

Expected results: Improved DLB diagnosis performance using a combination of multimodal biomarkers (EEG, cognitive scores, plasma, brain MRI).

ELIGIBILITY:
Inclusion Criteria for DLB ant AD patients:

* Neuropsychological assessment possible (good level in French language, absence of visual/auditory deficit limiting the cognitive assessment)
* Dementia with Lewy bodies according to the revised criteria of Mc Keith 2017 or probable AD defined according to McKhann 2011 criteria including CSF biomarkers (an abnormal level of beta-amyloid 1-42 protein [Ab42] or a pathological Ab42/Ab40 ratio and an abnormal level of phosphorylated tau [p-tau])

Inclusion Criteria for control patients:

* Neuropsychological assessment possible (good level in French language, absence of visual/auditory deficit limiting the cognitive assessment)
* MMSE (Mini-mental State Examination) greater than or equal to 28, normal MemScreen test results, normal brain MRI and normal neurological examination

Exclusion Criteria (for all) :

* Contraindication to MRI
* Other neurological or psychiatric or toxic/iatrogenic disorders that may account for the cognitive impairment or for EEG abnormalities
* Any unstable medical pathology and/or that may account for the cognitive impairment

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Observational prospective cohort study included at the GHU AP-HP. Nord Lariboisière, Cognitive Neurology Center : 50 probable DLB patients, 50 AD patients, and 30 control subjects with subjective cognitive impairment but without any element in favor of neurodegenerative disorders
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of a composite multimodal score | 24 month
  Diagnostic performance (sensitivity, specificity, accuracy) of a composite multimodal score combining quantitative EEG metrics, plasma biomarkers, MRI volumetric markers and cognitive scores, to differentiate groups of patients (AD, DLB) and control subjects.

SECONDARY OUTCOMES:
Comparison between groups of patients and controls of a composite EEG score combining several quantitative EEG parameters. | 24 month
Correlation between EEG parameters, biological biomarkers, MRI volumetric markers and cognitive scores assessed in the three groups (DLB, AD, controls) | 24 month
Reproducibility of 32-electrode EEG results with the 4 dry electrodes EEG cap | 24 month

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de neurologie Cognitive, Paris, France, France

IPD SHARING:
Plan to Share IPD: No